CLINICAL TRIAL: NCT05595980
Title: A Randomized, Parallel, Double-blind, Placebo-Controlled Study to Investigate the Effects of a Novel Probiotic on Gastrointestinal Health in Generally Healthy Adults
Brief Title: The Effects of a Novel Probiotic on Gastrointestinal Health in Generally Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BIO-CAT Microbials, LLC (Industry)
Collaborators: Biofortis Clinical Research, Inc. (Industry); Ohio State University (Other)
Responsible Party: Sponsor
Organization: BIO-CAT, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: BIO-2210
Record Dates: First submitted 2022-10-20; First posted 2022-10-27 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Gastrointestinal Health; Immune Health; Digestive Health
Keywords: Bacillus; probiotic; bloating; microbiome; metagenomics; inestinal; permeability
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Experimental): Bacillus strain spore preparation
  Interventions: Dietary Supplement: Probiotic
- Placebo (Placebo Comparator): Placebo maltodextrin
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — Participants will consume 1 capsule containing 2 billion CFU of a Bacillus strain spore preparation once daily for 56 days
  Arms: Probiotic
Dietary Supplement: Placebo — Participants will consume 1 capsule containing maltodextrin once daily for 56 days
  Arms: Placebo

SUMMARY:
The primary objective of this study is to investigate the effect of an oral probiotic (Bacillus sp. spore preparation) on abdominal bloating, flatulence, and burping in generally healthy adults. Secondary outcomes include intestinal barrier integrity and fecal microbiome properties (taxonomical structure, diversity, and function).

DETAILED DESCRIPTION:
Probiotics are live microbes that, when administered in adequate amounts, confer a health benefit. Examples of probiotic health benefits include the support of gastrointestinal (GI) health and immune health. Common probiotic strains include species from the Bacillaceae family (e.g. Bacillus genus) and Lactobacillaceae family of the Bacillota phylum (formerly Firmicutes), and species from the Bifidobacterium genus of the Actinomycetota phylum (formerly Actinobacteria). Bacillaceae species are particularly advantageous for oral probiotic applications because they can be manufactured as spores with highly proteinaceous coats that persist without refrigeration and resist the acidic and high bile salt conditions that occur across the human GI tract. The objective of this clinical study is to investigate the effects of daily oral supplementation with a novel Bacillus sp. spore preparation for 8 weeks on GI symptoms, intestinal barrier integrity, and fecal microbiome properties.

This will be a randomized, parallel, double-blind, placebo-controlled study consisting of one screening visit (Visit 1, Day -7) and four study visits (Days 0, 1, 57, and 58). At Visit 1 (Day -7), participants will arrive at the clinic in a fasting state (≥ 10 hours). After participants provide voluntary informed consent, participants will undergo medical history, prior and current medication/supplement use, and inclusion and exclusion criteria assessments. Additionally, height, body weight, and vital signs will be measured, and body mass index (BMI) will be calculated. Blood samples will be collected for chemistry, hematology, C-reactive protein (CRP), and insulin analyses. Participants will be dispensed a daily paper Gastrointestinal Tolerance Questionnaire (GITQ) with instructions to capture events occurring during the seven continuous days prior to Visit 2 (Day 0). The paper GITQ contains a series of questions regarding the presence and severity of GI symptoms occurring during the past 24 hours. Therefore, participants will be instructed to complete their first GITQ on the morning of Day -6 and the final GITQ on the morning of Day 0, just before their Visit 2. Additionally, a stool sample collection kit will be dispensed with instructions to a collect stool sample from a single bowel movement (for fecal microbiome analyses) within the 3 days immediately before Visit 2 (Day 0).

At Visit 2 (Day 0), participants will arrive at the clinic in a fasting state (≥ 10 hours). Participants will undergo clinic visit procedures (concomitant medication/supplement use, assess inclusion/exclusion criteria, body weight, and vital signs measurements) and adverse event (AE) assessment. Fecal samples will be collected, and subjects will be administered a 7-day recall GITQ. Participants will then undergo an intestinal permeability test where they will ingest four sugar probes (1 g mannitol, 1 g sucralose, 1 g erythritol, and 5 g lactulose) in approximately 240 mL water. Participants will be dispensed 2 separate containers to collect all urine over the following 24 hours, with urine collected from 0 to 5 hours in one container and from 5 to 24 hours in the second container. Participants will be instructed to return both containers to the clinic the following day at Visit 3 (Day 1). Upon completion of the GI permeability test, participants will be randomly assigned to a study product sequence. Participants will receive an email link for an electronic 7-day recall GITQ to be completed on Days 8, 15, 22, 29, 36, 43, 50, and 57. Participants will also receive information regarding daily links that will be sent via email to complete electronic 24-hour recall GITQs and will be instructed to complete these electronic 24-hour GITQs daily starting on day 51, which will be 6 days ahead of Visit 4. Participants will continue recording the 24-hour GITQ recall every day for seven total days (Days 51, 52, 53, 54, 55, 56, and 57). Additionally, a stool sample collection kit will be dispensed with instructions to collect a stool sample from a single bowel movement for fecal microbiome analyses within the 3 days immediately before Visit 4 (Day 57). In addition, a subset of male subjects will be selected to collect an additional fecal sample for fecal metabolomic and/or targeted analyte analyses.

At Visit 3 (Day 1), participants will return the 24-hour urine sample collection containers and undergo AE assessments. Participants will be dispensed their assigned study product and will be instructed to consume it once a day (1 capsule/d) with their meal that is typically the largest of the day for 56 days starting on Day 1.

At Visit 4 (Day 57), participants will arrive at the clinic fasted (≥ 10 hours) and undergo clinic visit procedures, including: concomitant medication/supplement use, review inclusion/exclusion criteria, body weight and vital signs measurements, and AE assessment. Fecal samples will be collected. Blood samples will be collected for chemistry, hematology, CRP, and insulin analyses. Participants will then complete the intestinal permeability test with the same procedures and study instructions described at Visit 2.

At Visit 5 (Day 58), participants will return the 24-hour urine sample collection containers and undergo AE assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 30-65 years of age, inclusive at Visit 1 (Day -7)
2. BMI of 18.50 to 31.99 kg/m^2, inclusive, at Visit 1 (Day -7)
3. Have ≥ 3 weekly total symptom score obtained by combining ratings for gas/flatulence, abdominal bloating, and burping symptoms (e.g., 3 days with a mild severity across the three symptoms, 1 day of mild severity and 1 day of moderate severity across the three symptoms, or 1 day of severe severity across the three symptoms)
4. Consumes a typical American diet (defined as ≤ 3 servings/d of fruits and vegetables combined and < 3 servings/d of whole grains)
5. Non-user of tobacco or nicotine products (e.g., cigarette smoking, vaping, chewing tobacco) with no plans to begin use during the study period
6. Non-user or former users (cessation ≥ 12 months) of any marijuana or hemp products and has no plans to use marijuana or hemp products during the study period
7. Willing to maintain physical activity and exercise patterns, body weight, and habitual diet throughout the trial
8. Willing to limit alcohol consumption to ≤ 2 standard drinks per day throughout the trial
9. Willing to refrain from exclusionary medications, supplements, and products throughout the study
10. No health conditions that would prevent him/her from fulfilling the study requirements as judged by the Clinical Investigator on the basis of medical history and routine laboratory test results
11. Understands the study procedures and signs forms providing informed consent to participate in the study and authorizes the release of relevant protected health information to the Clinical Investigator

Exclusion Criteria:

1. Known sensitivity, intolerability, or allergy to any of the study products or their excipients
2. Abnormal laboratory test results of clinical significance at Visit 1 (Day -7), at the discretion of the Clinical Investigator
3. Clinically important GI condition that would potentially interfere with the evaluation of the study product (e.g., inflammatory bowel disease, irritable bowel syndrome, gastric reflux, indigestion, dyspepsia, Crohn's disease, celiac disease, history of surgery for weight loss, gastroparesis, and clinically significant lactose or gluten intolerance or other food or ingredient allergies)
4. Pre-menopausal female subject with an irregular menstrual cycle (regular cycle defined as 21 to 35 days in length for the last 3 months prior to Visit 1)
5. Recent (within 2 weeks of Visit 1; Day -7) history of an episode of acute GI illness such as nausea/vomiting or diarrhea (defined as ≥ 3 loose or liquid stools/d)
6. Self-reported history (within 6 weeks of Visit 1; Day -7) of constipation (defined as fewer than three bowel movements per week)
7. Uncontrolled and/or clinically important pulmonary (including uncontrolled asthma), cardiac (including, but not limited to, atherosclerotic disease, history of myocardial infarction, peripheral arterial disease, stroke), hepatic, renal, endocrine (including Type 1 and Type 2 diabetes mellitus), hematologic, immunologic, neurologic (such as Alzheimer's or Parkinson's disease), psychiatric (including depression and/or anxiety disorders) or biliary disorders. Conditions which are well-controlled or resolved will be assessed by the Clinical Investigator on a case-by-case basis.
8. Uncontrolled hypertension (systolic blood pressure ≥ 140 mm Hg or diastolic blood pressure ≥ 90 mm Hg) as defined by the blood pressure measured at Visit 1 (Day -7)
9. Have received a COVID-19 vaccine within 2 weeks of randomization or expected to receive a COVID-19 vaccine during the study period
10. Had a positive SARS-CoV2 test and experienced symptoms for > 2 months (i.e. "long-haulers")
11. Known allergy, intolerances or sensitivity to milk, soy, or wheat
12. Extreme dietary habits at the discretion of the Clinical Investigator
13. History or presence of cancer in the prior 2 years, except for non-melanoma skin cancer
14. Major trauma or any other surgical event within 3 months of Visit 1 (Day -7)
15. Signs or symptoms of an active infection of clinical relevance within 5 days of Visit 1 (Day -7)
16. Weight loss or gain > 4.5 kg in the 3 months prior to Visit 1 (Day -7)
17. Currently or planning to be on a weight loss regimen during the study
18. Antibiotic use within 3 months of Visit 1 (Day -7) and throughout the study period
19. Use of steroids within 1 month of Visit 1 (Day -7) and throughout the study period
20. Chronic use (i.e., daily on a regular basis) of anti-inflammatory medications (e.g., NSAIDS) within 1 month of Visit 1 (Day -7)
21. Use of medications (over-the-counter or prescription) and/or dietary supplements, known to influence GI function, including but not limited to, pre- and probiotic supplements as well as foods or beverages containing live probiotics (e.g., yogurt, kombucha), fiber supplements, laxatives, enemas, suppositories, H2 blockers, proton pump inhibitors, antacids, anti-diarrheal agents, anti-depressants, and/or anti-spasmodic within 2 weeks of Visit 1 (Day -7) and throughout the study period
22. Participated in endoscopy or endoscopy preparation within 3 months prior to Visit 1 (Day -7)
23. Exposure to any non-registered drug product within 4 weeks prior to Visit 1 (Day -7)
24. Female who is pregnant, planning to be pregnant during the study period, lactating, or is of childbearing potential and is unwilling to commit to the use of a medically approved form of contraception throughout the study period
25. Recent history (within 12 months of screening; Visit 1; Day -7) of alcohol or substance abuse
26. Self-report of blood donation totaling between 101 mL to 449 mL of blood within 30 days prior to screening or a blood donation of more than 450 mL within 56 days
27. Receipt or use of study products in another research study within 28 days prior to Visit 2 (Day 0) or longer if the previous study product is deemed by the Clinical Investigator to have lasting effects that might influence the eligibility criteria or outcomes of current study.
28. Has a condition the Clinical Investigator believes would interfere with his ability to provide informed consent, comply with the study protocol, which might confound the interpretation of the study results, or put the subject at undue risk

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-09-19 (Actual); Primary Completion 2023-02-03 (Actual); Study Completion 2023-02-03 (Actual)

PRIMARY OUTCOMES:
Composite score of abdominal bloating, flatulence, and burping (daily GITQ) | 9 weeks
  Between placebo and probiotic treatments, the difference in the proportion of participants with a decrease (indicating improvement) in the 7-day total composite score of abdominal bloating, flatulence, and burping, from baseline to week 8, where an increase in scores (indicating worsening) cannot occur within any of the 3 symptoms (daily Gastrointestinal Tolerance Questionnaire [GITQ])

SECONDARY OUTCOMES:
Composite score of abdominal bloating, flatulence, and burping (7-day recall GITQ) | 9 weeks
  Between placebo and probiotic treatments, the difference in the proportion of participants with a decrease in the 7-day total composite score of abdominal bloating, flatulence, and burping, from baseline to week 8 (7-day recall GITQ)
Composite score of 8 GI symptoms (daily GITQ) | 9 weeks
  Between placebo and probiotic treatments, the difference in the proportion of participants with a decrease in the 7-day total composite score of abdominal bloating, flatulence, burping, nausea, vomiting, abdominal cramping, stomach rumbling, and reflux, from baseline to week 8 (daily GITQ)
Composite score of 8 GI symptoms (7-day recall GITQ) | 9 weeks
  Between placebo and probiotic treatments, the difference in the proportion of participants with a decrease in the 7-day total composite score of abdominal bloating, flatulence, burping, nausea, vomiting, abdominal cramping, stomach rumbling, and reflux, from baseline to week 8 (7-day recall GITQ)
Individual GI symptom scores (daily GITQ) | 9 weeks
  Between placebo and probiotic treatments, the difference in the proportion of participants with a decrease in 7-day individual symptom scores from baseline to week 8, for each of abdominal bloating, flatulence, burping, nausea, vomiting, abdominal cramping, stomach rumbling, and reflux (daily GITQ)
Individual GI symptom scores (7-day recall GITQ) | 9 weeks
  Between placebo and probiotic treatments, the difference in the proportion of participants with a decrease in 7-day individual symptom scores from baseline to week 8, for each of abdominal bloating, flatulence, burping, nausea, vomiting, abdominal cramping, stomach rumbling, and reflux (7-day recall GITQ)
Composite score of abdominal bloating, flatulence, and burping (interim weeks) | 2 - 8 weeks
  Between placebo and probiotic treatments, the difference in the proportion of participants showing a decrease in the 7-day total composite score of abdominal bloating, flatulence, and burping, from baseline to each measured, interim time point (i.e., week 1, week 2, week 3, week 4, week 5, week 6, week 7) (7-day recall GITQ)
Individual GI symptom scores (interim weeks) | 2 - 8 weeks
  Between placebo and probiotic treatments, the difference in the proportion of participants showing a decrease in the 7-day individual symptom scores for each of abdominal bloating, flatulence, burping, nausea, vomiting, abdominal cramping, stomach rumbling, and reflux, from baseline to each measured, interim time point (i.e., week 1, week 2, week 3, week 4, week 5, week 6, week 7) (7-day recall GITQ)
Small intestinal permeability | 8 weeks
  Between placebo and probiotic treatments, the difference in small intestinal permeability from baseline to Day 57 (0 to 5 hour urinary lactulose:mannitol ratio)
Colonic permeability | 8 weeks
  Between placebo and probiotic treatments, the difference in colonic permeability from baseline to Day 57 (5 to 24 hour urinary sucralose:erythritol ratio)
Gut permeability | 8 weeks
  Between placebo and probiotic treatments, the difference in gut permeability from baseline to Day 57 (0 to 24 hour urinary sucralose:erythritol ratio)
Fecal microbiome profile | 8 weeks
  Between placebo and probiotic treatments, the difference in "shotgun" metagenomic sequencing-based fecal microbiome profiles from baseline to Day 57
Fecal microbiome profile | Day 57
  Between placebo and probiotic treatments, the difference in "shotgun" metagenomic sequencing-based fecal microbiome profiles at end of study
Plasma C-reactive protein | 9 weeks
  Between placebo and probiotic treatments, change from baseline to week 8 in fasting blood C-reactive protein concentration (mg/L)
Serum insulin | 9 weeks
  Between placebo and probiotic treatments, change from baseline to week 8 in fasting serum insulin concentration (mIU/L)
Safety: Albumin | 9 weeks
  Fasting plasma albumin concentration (g/dL)
Safety: Alkaline phosphatase | 9 weeks
  Fasting plasma alkaline phosphatase concentration (U/L)
Safety: Alanine aminotransferase | 9 weeks
  Fasting plasma alanine aminotransferase concentration (U/L)
Safety: Anion gap | 9 weeks
  Fasting plasma anion gap (nmol/L)
Safety: Aspartate aminotransferase | 9 weeks
  Fasting plasma aspartate aminotransferase concentration (U/L)
Safety: Blood urea nitrogen | 9 weeks
  Fasting blood urea nitrogen concentration (mg/dL)
Safety: Osmolality | 9 weeks
  Fasting plasma osmolality (mOsm/kg)
Safety: Calcium | 9 weeks
  Fasting plasma total calcium concentration (mg/dL)
Safety: Chloride | 9 weeks
  Fasting plasma chloride concentration (mmol/L)
Safety: Carbon dioxide | 9 weeks
  Fasting plasma carbon dioxide concentration (mmol/L)
Safety: Creatinine | 9 weeks
  Fasting plasma creatinine concentration (mg/dL)
Safety: Globulin | 9 weeks
  Fasting plasma globulin concentration (g/dL)
Safety: Glucose | 9 weeks
  Fasting plasma glucose concentration (mg/dL)
Safety: Potassium | 9 weeks
  Fasting plasma potassium concentration (mmol/L)
Safety: Sodium | 9 weeks
  Fasting plasma sodium concentration (mmol/L)
Safety: Total bilirubin | 9 weeks
  Fasting plasma total bilirubin concentration (mg/dL)
Safety: Total protein | 9 weeks
  Fasting plasma total protein concentration (g/dL)
Safety: Basophils | 9 weeks
  Fasting plasma basophil count
Safety: Eosinophils | 9 weeks
  Fasting plasma eosinophil count
Safety: Hematocrit | 9 weeks
  Fasting hematocrit (as volume percent)
Safety: Hemoglobin | 9 weeks
  Fasting plasma hemoglobin concentration (g/dL)
Safety: Lymphocytes | 9 weeks
  Fasting plasma lymphocyte count
Safety: Mean corpuscular hemoglobin | 9 weeks
  Fasting plasma mean corpuscular hemoglobin (pg)
Safety: Mean corpuscular hemoglobin concentration | 9 weeks
  Fasting plasma mean corpuscular hemoglobin concentration (g/dL)
Safety: Mean corpuscular volume | 9 weeks
  Fasting plasma mean corpuscular volume (fL)
Safety: Monocytes | 9 weeks
  Fasting plasma monocyte count
Safety: Neutrophils | 9 weeks
  Fasting plasma neutrophil count
Safety: Platelets | 9 weeks
  Fasting plasma platelet count
Safety: Red blood cells | 9 weeks
  Fasting plasma red blood cell count
Safety: White blood cells | 9 weeks
  Fasting plasma white blood cell count
Safety: Blood pressure | 9 weeks
  Resting systolic blood pressure over resting diastolic blood pressure (mmHg/mmHg)
Safety: Heart rate | 9 weeks
  Resting heart rate (beats per minute)
Safety: Incidence of adverse events | 9 weeks
  Number of participants with self-reported adverse events

OTHER OUTCOMES:
Fecal metabolome profile | Day 57
  Between placebo and probiotic treatments, the difference in the mass spectrometry-based fecal metabolome profiles at end of study (only for 16 to 20 male participants with BMI 25.00-31.99 kg/(m)^2)

CONTACTS AND LOCATIONS:
Overall Officials: Dawn Beckman, MD, Principal Investigator — Biofortis Clinical Research, Inc.
Locations (1):
- Biofortis Clinical Research, Inc., Addison, Illinois, United States

IPD SHARING:
Plan to Share IPD: No